CLINICAL TRIAL: NCT02781129
Title: Memory, Epilepsy and Brain Stimulation: Oscillatory Patterns During Real-world Navigation and Free Recall in Chronically Implanted Humans
Brief Title: Navigation and Free Recall in Chronically Implanted Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Jobst (Other)
Collaborators: NeuroPace (Industry)
Responsible Party: Sponsor-Investigator, Barbara Jobst, Dr., Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D16119
Record Dates: First submitted 2016-05-05; First posted 2016-05-24 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy
Keywords: Memory; Responsive Neurostimulator System
MeSH Terms: conditions — Epilepsy | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RNS® Neurostimulator (Experimental): Subjects with pharmaceutically intractable seizures who have been implanted with a RNS® Neurostimulator.
  Interventions: Other: electrical stimulation

INTERVENTIONS:
Other: electrical stimulation — Stimulation applied will be within parameters commonly used for the treatment of epilepsy during periods of encoding, recall, and memory maintenance .

SUMMARY:
This study is designed to identify brain activity associated with good memory in subjects with a chronically implanted RNS® device and to study the effects of therapeutic stimulation for epilepsy on memory. This will be accomplished through analysis of ECoG data collected during memory encoding for short and long-term free recall as well as during navigation tasks.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent
* 18 years of age or older
* Diagnosis of epilepsy
* Implanted RNS® device and receiving therapeutic stimulation for epilepsy.
* Capable of completing experimental tasks in the judgment of the Principal Investigator

Exclusion Criteria:

* RNS® Neurostimulator implanted within 3 months of experimental tasks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2025-05 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
Proportion of words recalled with and without stimulation. | 30 days
  This study is designed to study the effects of therapeutic stimulation for epilepsy on memory. This outcome will be assessed by free recall language and memory tasks.

SECONDARY OUTCOMES:
Changes in the power spectrum of ECoG data with an increase of recalled words. | 30 days
  This study is designed to identify brain activity associated with good memory in subjects with a chronically implanted RNS® device. This outcome will be assessed by free recall language and memory tasks.
Proportion of words recalled during times of interictal activity. | 30 days
  This study is designed to investigate the effects of IEDs on spatial, long-term, and short-term memory. This will be assessed by free recall language and memory tasks.
Proportion of navigation challenges recalled successfully with and without stimulation. | 30 days
  This outcome will be assessed by real-world and virtual navigation tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara C Jobst, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center in Lebanon, NH, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No